CLINICAL TRIAL: NCT02843191
Title: KCSP Trial of CONsolidation Chemotherapy for Locally Advanced Mid or Low Rectal Cancer After NeoadjUvant Concurrent ChemoraDiothErapy: a Multicenter, Randomized Controlled Trial (KONCLUDE)
Brief Title: Consolidation Chemotherapy for Locally Advanced Mid or Low Rectal Cancer After Neoadjuvant Concurrent Chemoradiotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Korean Society of ColoProctology (Unknown); Pharmbio Korea Inc. (Unknown); Samjin Pharmaceutical Co., Ltd. (Industry); Boryung Pharmaceutical Co., Ltd (Industry); JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Suk-Hwan Lee, Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSCP2016
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Consolidation Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Adjuvant chemotherapy (Active Comparator): After neoadjuvant chemoradiotherapy, patients will receive surgery followed by eight cycles of chemotherapy.
  Interventions: Drug: Chemotherapy
- Consolidation chemotherapy (Experimental): After neoadjuvant chemoradiotherapy, patients will receive three cycles of chemotherapy. Thereafter, they will receive surgery followed by five cycles of chemotherapy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — 5-FU, Leucovorin, and Oxaliplatin (FOLFOX regimen)

SUMMARY:
This trial is to assess the efficacy and feasibility of consolidation chemotherapy after neoadjuvant chemoradiotherapy for locally advanced mid or low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of mid or low rectum
2. Locally advanced rectal cancer confirmed by image (i.e. Magnetic resonance image)

   * Clinical stage T1-3N1or2 on MRI
   * Clinical stage cT3N0 (or depth of perirectal invasion by tumor >5mm on MRI)
   * Suspicious of circumferential invasion on MRI (or circumferential margin <1mm)
3. ECOG performance status of 0-2
4. ASA grade ≤ 3
5. An informed consent has been signed by the patient

Exclusion Criteria:

1. Upper rectal cancer
2. Clinical stage T1or2N0 on MRI
3. Clinical stage T4Nany on MRI
4. Clinical stage TanyNanyM1 by image or histology
5. The patient received chemotherapy or radiotherapy during the past 6 months
6. The patient received any therapy for colorectal cancer or another malignancy during the past 5 years
7. The patient has severe underlying diseases or poor condition to receive chemotherapy or radiotherapy
8. Pregnant of breastfeeding women
9. The patient who participate in another clinical trial, or receives any drug for the trial
10. Uncontrolled peripheral neuropathy (more than grade 2)
11. Any unhealed wound, fracture, peptic ulcer, or intraabdominal abscess
12. Active gastrointestinal bleeding
13. Patients with an active infection, which needs antibiotic therapy, during the randomization period

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 2 years
  Pathologic complete response is defined as no residual tumor on the surgical specimen after chemoradiotherapy. (i.e. Mandard grade 1 or Dworak grade 4)
Disease-free survival | 3 years
  The rates of patients who survive without recurrence

SECONDARY OUTCOMES:
Radiotherapy-related complications | 2 years
  Complications according to the CTCAE 4.0
R0 resection | 2 years
  R0 resection is defined as resection without remnant tumor, whereas R1 resection as microscopic residual tumor and R2 resection as gross residual tumor. R0 resection will be proven histologically as no resection margin involvement of tumor.
Tumor response rate | 2 years
  Amount of tumor regression after surgery according to the guideline including Mandard or Dworak
Postoperative complications | 2 years
  Complications after surgery
Peripheral neuropathy | 3 years
  Peripheral neuropathy will be evaluated as grade 1 to 4 according to NCI CTCAE 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Hwan Lee, MD, PhD, Principal Investigator — 892 Dongnam-ro, Gangdong-gu, Seoul, Korea. Kyung Hee University Hospital at Gangdong; Chang Woo Kim, MD, PhD, Study Director — 164 Worldcup-ro, Yeongtong-gu, Suwon, Korea. Ajou University School of Medicine
Locations (14):
- South Korea (14):
  - Inje University Busan Paik hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chuncheon Sacred Heart Hospital, Hallym University College of Medicine, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Wonkwang University Hospital, Iksan
  - Inje University Sanggye Paik Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul
  - Seoul St. Mary's Hospital, The Catholic University College of Medicine, Seoul
  - Ajou University School of Medicine, Suwon
  - Uijeongbu St. Mary's Hospital, The Catholic University College of Medicine, Uijeongbu-si
  - Wonju Severance Christian Hospital, Yonsei University Wonju College of Medicine, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Kapiteijn E, Kranenbarg EK, Steup WH, Taat CW, Rutten HJ, Wiggers T, van Krieken JH, Hermans J, Leer JW, van de Velde CJ. Total mesorectal excision (TME) with or without preoperative radiotherapy in the treatment of primary rectal cancer. Prospective randomised trial with standard operative and histopathological techniques. Dutch ColoRectal Cancer Group. Eur J Surg. 1999 May;165(5):410-20. doi: 10.1080/110241599750006613. PMID 10391155
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Gastrointestinal Tumor Study Group. Prolongation of the disease-free interval in surgically treated rectal carcinoma. N Engl J Med. 1985 Jun 6;312(23):1465-72. doi: 10.1056/NEJM198506063122301. PMID 2859523
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Roh MS, Colangelo LH, O'Connell MJ, Yothers G, Deutsch M, Allegra CJ, Kahlenberg MS, Baez-Diaz L, Ursiny CS, Petrelli NJ, Wolmark N. Preoperative multimodality therapy improves disease-free survival in patients with carcinoma of the rectum: NSABP R-03. J Clin Oncol. 2009 Nov 1;27(31):5124-30. doi: 10.1200/JCO.2009.22.0467. Epub 2009 Sep 21. PMID 19770376
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Valentini V, Coco C, Picciocchi A, Morganti AG, Trodella L, Ciabattoni A, Cellini F, Barbaro B, Cogliandolo S, Nuzzo G, Doglietto GB, Ambesi-Impiombato F, Cosimelli M. Does downstaging predict improved outcome after preoperative chemoradiation for extraperitoneal locally advanced rectal cancer? A long-term analysis of 165 patients. Int J Radiat Oncol Biol Phys. 2002 Jul 1;53(3):664-74. doi: 10.1016/s0360-3016(02)02764-5. PMID 12062610
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976
- [Background] Mandard AM, Dalibard F, Mandard JC, Marnay J, Henry-Amar M, Petiot JF, Roussel A, Jacob JH, Segol P, Samama G, et al. Pathologic assessment of tumor regression after preoperative chemoradiotherapy of esophageal carcinoma. Clinicopathologic correlations. Cancer. 1994 Jun 1;73(11):2680-6. doi: 10.1002/1097-0142(19940601)73:113.0.co;2-c. PMID 8194005
- [Background] Garcia-Aguilar J, Hernandez de Anda E, Sirivongs P, Lee SH, Madoff RD, Rothenberger DA. A pathologic complete response to preoperative chemoradiation is associated with lower local recurrence and improved survival in rectal cancer patients treated by mesorectal excision. Dis Colon Rectum. 2003 Mar;46(3):298-304. doi: 10.1007/s10350-004-6545-x. PMID 12626903
- [Background] Dworak O, Keilholz L, Hoffmann A. Pathological features of rectal cancer after preoperative radiochemotherapy. Int J Colorectal Dis. 1997;12(1):19-23. doi: 10.1007/s003840050072. PMID 9112145
- [Background] Gerard JP, Azria D, Gourgou-Bourgade S, Martel-Laffay I, Hennequin C, Etienne PL, Vendrely V, Francois E, de La Roche G, Bouche O, Mirabel X, Denis B, Mineur L, Berdah JF, Mahe MA, Becouarn Y, Dupuis O, Lledo G, Montoto-Grillot C, Conroy T. Comparison of two neoadjuvant chemoradiotherapy regimens for locally advanced rectal cancer: results of the phase III trial ACCORD 12/0405-Prodige 2. J Clin Oncol. 2010 Apr 1;28(10):1638-44. doi: 10.1200/JCO.2009.25.8376. Epub 2010 Mar 1. PMID 20194850
- [Background] Aschele C, Cionini L, Lonardi S, Pinto C, Cordio S, Rosati G, Artale S, Tagliagambe A, Ambrosini G, Rosetti P, Bonetti A, Negru ME, Tronconi MC, Luppi G, Silvano G, Corsi DC, Bochicchio AM, Chiaulon G, Gallo M, Boni L. Primary tumor response to preoperative chemoradiation with or without oxaliplatin in locally advanced rectal cancer: pathologic results of the STAR-01 randomized phase III trial. J Clin Oncol. 2011 Jul 10;29(20):2773-80. doi: 10.1200/JCO.2010.34.4911. Epub 2011 May 23. PMID 21606427
- [Background] Gerard JP, Azria D, Gourgou-Bourgade S, Martel-Lafay I, Hennequin C, Etienne PL, Vendrely V, Francois E, de La Roche G, Bouche O, Mirabel X, Denis B, Mineur L, Berdah JF, Mahe MA, Becouarn Y, Dupuis O, Lledo G, Seitz JF, Bedenne L, Juzyna B, Conroy T. Clinical outcome of the ACCORD 12/0405 PRODIGE 2 randomized trial in rectal cancer. J Clin Oncol. 2012 Dec 20;30(36):4558-65. doi: 10.1200/JCO.2012.42.8771. Epub 2012 Oct 29. PMID 23109696
- [Background] Bujko K, Nowacki MP, Nasierowska-Guttmejer A, Michalski W, Bebenek M, Kryj M. Long-term results of a randomized trial comparing preoperative short-course radiotherapy with preoperative conventionally fractionated chemoradiation for rectal cancer. Br J Surg. 2006 Oct;93(10):1215-23. doi: 10.1002/bjs.5506. PMID 16983741
- [Background] Ngan SY, Burmeister B, Fisher RJ, Solomon M, Goldstein D, Joseph D, Ackland SP, Schache D, McClure B, McLachlan SA, McKendrick J, Leong T, Hartopeanu C, Zalcberg J, Mackay J. Randomized trial of short-course radiotherapy versus long-course chemoradiation comparing rates of local recurrence in patients with T3 rectal cancer: Trans-Tasman Radiation Oncology Group trial 01.04. J Clin Oncol. 2012 Nov 1;30(31):3827-33. doi: 10.1200/JCO.2012.42.9597. Epub 2012 Sep 24. PMID 23008301
- [Background] Garcia-Aguilar J, Smith DD, Avila K, Bergsland EK, Chu P, Krieg RM; Timing of Rectal Cancer Response to Chemoradiation Consortium. Optimal timing of surgery after chemoradiation for advanced rectal cancer: preliminary results of a multicenter, nonrandomized phase II prospective trial. Ann Surg. 2011 Jul;254(1):97-102. doi: 10.1097/SLA.0b013e3182196e1f. PMID 21494121
- [Background] Gao YH, Lin JZ, An X, Luo JL, Cai MY, Cai PQ, Kong LH, Liu GC, Tang JH, Chen G, Pan ZZ, Ding PR. Neoadjuvant sandwich treatment with oxaliplatin and capecitabine administered prior to, concurrently with, and following radiation therapy in locally advanced rectal cancer: a prospective phase 2 trial. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1153-60. doi: 10.1016/j.ijrobp.2014.07.021. Epub 2014 Oct 13. PMID 25442042
- [Background] Nilsson PJ, van Etten B, Hospers GA, Pahlman L, van de Velde CJ, Beets-Tan RG, Blomqvist L, Beukema JC, Kapiteijn E, Marijnen CA, Nagtegaal ID, Wiggers T, Glimelius B. Short-course radiotherapy followed by neo-adjuvant chemotherapy in locally advanced rectal cancer--the RAPIDO trial. BMC Cancer. 2013 Jun 7;13:279. doi: 10.1186/1471-2407-13-279. PMID 23742033
- [Background] Hong YS, Nam BH, Kim KP, Kim JE, Park SJ, Park YS, Park JO, Kim SY, Kim TY, Kim JH, Ahn JB, Lim SB, Yu CS, Kim JC, Yun SH, Kim JH, Park JH, Park HC, Jung KH, Kim TW. Oxaliplatin, fluorouracil, and leucovorin versus fluorouracil and leucovorin as adjuvant chemotherapy for locally advanced rectal cancer after preoperative chemoradiotherapy (ADORE): an open-label, multicentre, phase 2, randomised controlled trial. Lancet Oncol. 2014 Oct;15(11):1245-53. doi: 10.1016/S1470-2045(14)70377-8. Epub 2014 Sep 4. PMID 25201358
- [Background] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Derived] Kim CW, Kang BM, Kim IY, Kim JY, Park SJ, Park WC, Bae KB, Bae BN, Baek SK, Baik SH, Son GM, Lee YS, Lee SH. Korean Society of Coloproctology (KSCP) trial of cONsolidation Chemotherapy for Locally advanced mid or low rectal cancer after neoadjUvant concurrent chemoraDiothErapy: a multicenter, randomized controlled trial (KONCLUDE). BMC Cancer. 2018 May 8;18(1):538. doi: 10.1186/s12885-018-4466-7. PMID 29739356